CLINICAL TRIAL: NCT07353528
Title: Development and Validation of a Machine Learning Model to Predict Hypothermia in Gynecological Laparoscopic Surgery Based on Preoperative Clinical Indicators: A Multicenter Prospective Cohort Study
Brief Title: Predicting Hypothermia in Gynecological Laparoscopic Surgery Using Machine Learning
Status: Not yet recruiting | Type: Observational
Sponsor: Chengdu Jinjiang Maternity and Child Health Hospital (Other)
Collaborators: Sichuan Jinxin Xinan Women & Children's Hospital (Unknown); People ' s Hospital of Dayi County (Unknown); Medical Center Hospital of QiongLai City (Unknown)
Responsible Party: Principal Investigator, Fei Jia, Director of Anesthesiology Department, Chengdu Jinjiang Maternity and Child Health Hospital
Other Study IDs: 202501
Record Dates: First submitted 2025-11-28; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Laparoscopic Surgery; Intraoperative Hypothermia; Gynecological Surgery
Keywords: Laparoscopic surgery; Intraoperative hypothermia; Machine learning; Gynecology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypothermia Group: This cohort consists of patients who develop intraoperative hypothermia (IOH) during gynecological laparoscopic surgery. IOH is defined as a core body temperature (measured by a wireless temperature monitoring system) falling below 36.0°C at any time during the surgery.
- Normothermia Group: This cohort comprises patients whose core body temperature (measured by a wireless temperature monitoring system) remains at or above 36.0°C throughout the entire gynecological laparoscopic surgery, and who do not develop intraoperative hypothermia (IOH). These patients serve as the control group for this study.

SUMMARY:
Brief Title: Predicting Hypothermia in Gynecological Laparoscopic Surgery Using Machine Learning

Brief Summary: This study aims to develop and validate a machine learning model for predicting intraoperative hypothermia (IOH) in patients undergoing gynecological laparoscopic surgery based on preoperative clinical indicators. This prospective, multicenter case-control study will enroll female patients aged 18 years and older who are scheduled for laparoscopic surgery across multiple hospitals from 2026 to 2027. The primary objective is to identify high-risk patients who may experience IOH, defined as a core temperature below 36.0°C during surgery.

Participants will be classified into two groups: the IOH group, consisting of patients who experience hypothermia, and the normal temperature group, comprising patients who maintain a core temperature of 36.0°C or higher. Data collection will include demographics, comorbidities, surgical details, anesthesia information, and preoperative laboratory results.

The primary outcome measure will be the area under the curve (AUC) of the model, assessing its predictive performance at various thresholds. Secondary outcomes will include sensitivity, positive predictive value, negative predictive value, and F1 score. The study hypothesizes that the developed machine learning model will significantly improve the accuracy and timeliness of predicting IOH, thereby enhancing patient safety during surgery and postoperative recovery. This research is expected to inform clinical practices related to preventative warming strategies, ultimately improving patient outcomes in gynecological laparoscopic surgery.

DETAILED DESCRIPTION:
Background: Intraoperative hypothermia (IOH), defined as a core body temperature below 36.0°C during surgery, is a common complication with an incidence as high as 50% in gynecological laparoscopic procedures. IOH is associated with adverse outcomes including surgical site infections, increased blood loss, cardiovascular complications, prolonged recovery, and higher healthcare costs. Accurate preoperative identification of patients at high risk for IOH is crucial for implementing targeted preventative measures and optimizing resource allocation.

Objective: The primary objective of this study is to develop and validate a machine learning model that utilizes preoperative clinical indicators to predict the occurrence of IOH specifically in patients undergoing gynecological laparoscopic surgery.

Study Design: This is a multicenter, prospective case-control study. Data will be prospectively collected from participating hospitals between 2026 and 2027.

Technical Methods:

Sample Size: Based on an estimated IOH incidence of 40% and 24 predictor variables, a minimum sample size of 1500 participants is planned to ensure adequate power for model development and validation.

Data Collection: Clinical data will be collected using electronic medical records (EMR). Core body temperature will be monitored intraoperatively using a wireless temperature monitoring system.

Statistical Analysis & Model Development: Data analysis will be performed using SPSS (v25.0) and R (v4.3.1). The dataset will be randomly split into training (80%) and testing (20%) sets. The Least Absolute Shrinkage and Selection Operator (LASSO) regression will be applied to the training set for feature selection. Six machine learning algorithms-Support Vector Machine (SVM), Logistic Regression (LR), Multilayer Perceptron (MLP), Random Forest (RF), Extreme Gradient Boosting (XGB), and Decision Tree (DT)-will be developed. Model hyperparameters will be optimized via 10-fold cross-validation.

Model Evaluation: The performance of all models will be independently validated on the test set. The primary metric for model comparison and selection will be the Area Under the Receiver Operating Characteristic Curve (AUC). Secondary performance metrics include sensitivity, positive predictive value (PPV), negative predictive value (NPV), and F1-score. The optimal cutoff point for the final selected model will be determined by maximizing Youden's index.

Ethical Considerations: This study will be conducted following approval by the Institutional Review Boards/Ethics Committees of all participating centers. Written informed consent will be obtained from all participants. The study protocol will be registered in a clinical trial registry to ensure transparency. All participant data will be handled with strict confidentiality and in accordance with relevant data protection regulations.

Expected Outcomes: This study is expected to result in a validated machine learning model capable of accurately predicting IOH risk prior to gynecological laparoscopic surgery. The identification of key predictive factors and the deployment of this model aim to facilitate personalized preventative care, reduce the incidence of IOH, and improve patient safety and postoperative recovery outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 years or older.
* Patients scheduled for laparoscopic surgery.

Exclusion Criteria:

* Preoperative body temperature exceeding 37.5°C or below 36.0°C.
* History of hypothyroidism or hyperthyroidism.
* Patients with thermoregulatory dysfunction, such as severe infection or central nervous system disorders.
* Patients who refuse to sign the informed consent form.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — eligibility is based on biological sex (female) as it pertains to the anatomical structures involved in the surgical procedure, not on gender identity.
Study Population: The study population consists of adult female patients undergoing gynecological laparoscopic surgery at multiple collaborating hospitals (including Chengdu Jinjiang District Maternal and Child Health Hospital, etc.). All participants must meet the inclusion criteria and not meet any exclusion criteria. Based on whether their intraoperative core temperature (measured by a wireless temperature monitoring system) falls below 36.0°C, patients will be categorized into either the "Hypothermia Group" (case) or the "Normothermia Group" (control). This is a prospective case-control study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Area Under the Receiver Operating Characteristic Curve (AUC) of the machine learning model for predicting intraoperative hypothermia | During surgery
  The primary outcome is the discriminatory performance of the developed machine learning model for predicting the occurrence of intraoperative hypothermia (defined as a core temperature < 36.0°C), as measured by the Area Under the Receiver Operating Characteristic Curve (AUC) evaluated on the independent testing set.

SECONDARY OUTCOMES:
Sensitivity | During surgery
  This metric measures the model's ability to correctly identify patients who will truly develop intraoperative hypothermia (true positive rate). It is calculated as the number of true positives divided by the sum of true positives and false negatives. This metric will be calculated on the model testing set.
Positive Predictive Value | During surgery
  This metric measures the proportion of patients predicted by the model to develop hypothermia who actually do so. It is calculated as the number of true positives divided by the sum of true positives and false positives. This metric will be calculated on the model testing set.
Negative Predictive Value | During surgery
  This metric measures the proportion of patients predicted by the model not to develop hypothermia who remain normothermic. It is calculated as the number of true negatives divided by the sum of true negatives and false negatives. This metric will be calculated on the model testing set.
F1-Score | During surgery
  This metric is the harmonic mean of precision (positive predictive value) and recall (sensitivity). It provides a single score that balances both concerns, especially useful when the class distribution is imbalanced. This metric will be calculated on the model testing set.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Chengdu Jinjiang District Women & Children Health Hospital, Chengdu, Sichuan
  - Sichuan Jinxin Xinan Women & Children's Hospital, Chengdu, Sichuan
  - People ' s Hospital of Dayi County, Chengdu, Sichuan
  - Medical Center Hospital of QiongLai City, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices) will be shared. Researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal will be granted access to the data. Proposals should be directed to the corresponding author via email. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Menzenbach J, Kirfel A, Guttenthaler V, Feggeler J, Hilbert T, Ricchiuto A, Staerk C, Mayr A, Coburn M, Wittmann M; PROPDESC Collaboration Group. PRe-Operative Prediction of postoperative DElirium by appropriate SCreening (PROPDESC) development and validation of a pragmatic POD risk screening score based on routine preoperative data. J Clin Anesth. 2022 Jun;78:110684. doi: 10.1016/j.jclinane.2022.110684. Epub 2022 Feb 18. PMID 35190344
- [Background] Lu Z, Chen X. Early prediction of intraoperative hypothermia in patients undergoing gynecological laparoscopic surgery: A retrospective cohort study. Medicine (Baltimore). 2024 Oct 4;103(40):e39038. doi: 10.1097/MD.0000000000039038. PMID 39465739
- [Background] Hosseini MP, Hosseini A, Ahi K. A Review on Machine Learning for EEG Signal Processing in Bioengineering. IEEE Rev Biomed Eng. 2021;14:204-218. doi: 10.1109/RBME.2020.2969915. Epub 2021 Jan 22. PMID 32011262
- [Background] Sessler DI, Pei L, Li K, Cui S, Chan MTV, Huang Y, Wu J, He X, Bajracharya GR, Rivas E, Lam CKM; PROTECT Investigators. Aggressive intraoperative warming versus routine thermal management during non-cardiac surgery (PROTECT): a multicentre, parallel group, superiority trial. Lancet. 2022 May 7;399(10337):1799-1808. doi: 10.1016/S0140-6736(22)00560-8. Epub 2022 Apr 4. PMID 35390321
- [Background] Cao B, Li Y, Liu Y, Chen X, Liu Y, Li Y, Wu Q, Ji F, Shu H. A multi-center study to predict the risk of intraoperative hypothermia in gynecological surgery patients using preoperative variables. Gynecol Oncol. 2024 Jun;185:156-164. doi: 10.1016/j.ygyno.2024.02.009. Epub 2024 Feb 29. PMID 38428331
- [Background] The nurse-nurse relationship. NLN Publ. 1990 Jun;(20-2294):257-61. No abstract available. PMID 2235395
- [Background] Gomez-Hidalgo NR, Pletnev A, Razumova Z, Bizzarri N, Selcuk I, Theofanakis C, Zalewski K, Nikolova T, Lanner M, Kacperczyk-Bartnik J, El Hajj H, Perez-Benavente A, Nelson G, Gil-Moreno A, Fotopoulou C, Sanchez-Iglesias JL. European Enhanced Recovery After Surgery (ERAS) gynecologic oncology survey: Status of ERAS protocol implementation across Europe. Int J Gynaecol Obstet. 2023 Jan;160(1):306-312. doi: 10.1002/ijgo.14386. Epub 2022 Aug 20. PMID 35929452
- [Background] Li L, Huang J, Chen X, Ma W, Hu Y, Li Y. A Retrospective Analysis of the Postoperative Effect of Intraoperative Hypothermia on Deep Vein Thrombosis After Intracranial Tumor Resection. World Neurosurg. 2022 Nov;167:e778-e783. doi: 10.1016/j.wneu.2022.08.099. Epub 2022 Aug 26. PMID 36038119
- [Background] Sessler DI. Perioperative thermoregulation and heat balance. Lancet. 2016 Jun 25;387(10038):2655-2664. doi: 10.1016/S0140-6736(15)00981-2. Epub 2016 Jan 8. PMID 26775126
- [Background] Carella M, Beck F, Piette N, Lecoq JP, Bonhomme VL. Effect of preoperative warming on intraoperative hypothermia and postoperative functional recovery in total hip arthroplasty: a randomized clinical trial. Minerva Anestesiol. 2024 Jan-Feb;90(1-2):41-50. doi: 10.23736/S0375-9393.23.17555-9. Epub 2023 Oct 25. PMID 37878246